CLINICAL TRIAL: NCT05509803
Title: Increasing Compliance With Physical Education Laws to Reduce Health Inequities
Brief Title: PE Audit and Feedback Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Hannah R. Thompson, Assistant Research Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1K01HL151805 (NIH)
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Physical Inactivity; Cardiovascular Diseases
MeSH Terms: conditions — Sedentary Behavior; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This will be a 2-group cluster-randomized clinical trial, with the school being the unit of assignment and randomization. 5 schools will receive an intervention and 5 schools will serve as controls.
Masking Description: This will be an intervention delivered at the school-level to improve physical education; blinding is not possible in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PE Audit and Feedback Intervention (Experimental): Schools in this arm will receive a PE audit and feedback tool delivered by the school district's teacher on special assignment for PE, which will consist of an audit of the school's existing PE program; Feedback on ways to improve the PE program; and technical assistance to help improve the PE program.
  Interventions: Behavioral: PE Audit and Feedback Tool
- PE Support as Usual (No Intervention): Schools in this arm will receive district-level support for PE as is typically provided by the school district.

INTERVENTIONS:
Behavioral: PE Audit and Feedback Tool — The intervention consists of a Physical Education (PE) Audit and Feedback tool, which was adapted from work done through the PE Works program in the New York City Department of Education. A district-level PE program leader in Oakland Unified School District will deliver the tool, which consists of auditing the current status of PE in intervention schools, providing feedback on the status to help improve PE, and providing technical assistance to bring schools up to code and ensure support for PE programming.
  Arms: PE Audit and Feedback Intervention

SUMMARY:
School physical education (PE) is one of the most valuable tools for increasing physical activity and fitness among youth of all backgrounds; however, compliance with existing PE laws is low (and differential by school race/ethnic and family-income composition, contributing to health disparities), and best practices for increasing compliance remain unknown. This study proposes to examine a novel approach for increasing PE law compliance by testing a PE audit and feedback tool (adapted from a tool used by the New York City Department of Education) in Oakland, California schools to determine the effectiveness, adaptability, and scalability of this potential cost-effective approach for increasing PE law compliance and student physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Elementary school in the Oakland Unified School District
* >50% of students in the school qualify for free or reduced-price meals
* >80% of students non-white

Exclusion Criteria:

* Having a PE program known by the PE Director to be well-established and/or meet/exceed district expectations for PE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness | Baseline (12 weeks); Follow-up (12 weeks)
  We will examine differences in changes between intervention and control schools from baseline in Fall 2020 to follow-up in Fall 2023 in 1) continuous estimated minutes of PE/week; and 2) binary meeting the California PE minute mandate of 200 minutes of PE/10 days for elementary students. We will calculate the estimated minutes of PE class-time students receive per week using the number of PE minutes scheduled per week, the proportion of scheduled PE classes that did not occur on days we randomly arrived to observe class, and actual observed PE class length from System for Observing Fitness Instruction Time (SOFIT) observations. Differences in changes in calculated minutes of PE/week and meeting the California PE minute mandate will be determined using adjusted linear and logistic mixed effects models with a time by group interaction term and random effects on teachers nested within school.
Adoption | 20-30 minutes
  To determine critical adoption issues, we will conduct 20-30 minute interviews with all observed teachers teaching PE and school principals after SOFIT observations are complete in the Fall of 2023. We will code all interview transcripts using a thematic analysis approach, using predefined themes based on the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) literature (e.g. commitment of principals and teachers; communication about the tool; impediments/facilitators to adoption, structural embedding of the tool into practice and policy, etc.).
Implementation | 20-30 minutes
  To determine critical implementation issues, we will conduct 20-30 minute interviews with all observed teachers teaching PE and school principals after SOFIT observations are complete in the Fall of 2023. We will code all interview transcripts using a thematic analysis approach, using predefined themes based on the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) literature (e.g. commitment of principals and teachers; communication about the tool; impediments/facilitators to implementation, structural embedding of the tool into practice and policy, etc.).
Maintenance | 20-30 minutes
  To determine critical maintenance issues, we will conduct 20-30 minute interviews with all observed teachers teaching PE and school principals after SOFIT observations are complete in the Fall of 2023. We will code all interview transcripts using a thematic analysis approach, using predefined themes based on the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) literature (e.g. commitment of principals and teachers; communication about the tool; impediments/facilitators to maintenance, structural embedding of the tool into practice and policy, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- UC Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No